CLINICAL TRIAL: NCT07291687
Title: Transcranial Direct Current Stimulation as a Treatment for Motor Function in Participants Living With Progressive Supranuclear Palsy, Corticalbasal Syndrome Degeneration, or Parkinson's Disease
Brief Title: tDCS as Treatment for Motor Function
Acronym: PSP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baycrest (Other)
Responsible Party: Principal Investigator, Tyler Roncero, Principle Investigator, Baycrest
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 21-17
Record Dates: First submitted 2025-11-17; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Progressive Supranuclear Palsy; Cortical Basal Ganglionic Degeneration; Parkinson Disease
Keywords: Progressive Supranuclear Palsy (PSP),; Cortical basal syndrome (CBD)
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The study is a Longitudinal A-B-A study with alternating between real (A) and sham sessions (B).
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS Stimulation: (Experimental): Participants will be exposed to 20 min of tDCS brain stimulation while undergoing training on cognitive tasks.
  Interventions: Device: Transcranial direct current stimulation (TDCS)
- Sham Arm (Placebo Comparator): Participants will be exposed to 20 min of tDCS sham/placebo stimulation while undergoing training on cognitive tasks. Participants will have the exact same apparatus used but with no stimulation.
  Interventions: Device: Stimulation Arm

INTERVENTIONS:
Device: Transcranial direct current stimulation (TDCS) — The Crossover design will enable us to use each participant as their own control.
  Arms: Real tDCS Stimulation:
Device: Stimulation Arm — Participants will be exposed to the brain stimulation protocol while undergoing certain motor task during the training sessions.
  Arms: Sham Arm

SUMMARY:
Previous preliminary results are sufficiently impressive to suggest that tDCS stimulation does have the potential to improve motor function when that ability is trained during stimulation. In the proposed study, the investigation will assess whether walking sessions combined with tDCS lead to improvements in motor function: gait, articulation, eye gaze, and motor dexterity. In addition, the investigators wish to examine if such results can be replicated in people with other conditions, such as cortical basal syndrome, and Parkinson's disease.

DETAILED DESCRIPTION:
Previous preliminary results are sufficiently impressive to suggest that tDCS stimulation does have the potential to improve motor function when that ability is trained during stimulation. In the proposed study, the investigators will assess whether walking sessions combined with tDCS lead to improvements in motor function: gait, articulation, eye gaze, and motor dexterity. In addition, the investigators wish to examine if such results can be replicated in people with other conditions, such as cortical basal syndrome, and Parkinson's disease. The rationale for including people living with these conditions is the overlap in motor and cortical network dysfunction observed across these disorders. All three conditions involve impairment of motor initiation, gait, coordination, and executive motor control due to degeneration in frontal-subcortical pathways. This extension will also allow for comparison of stimulation responsiveness across related diagnostic groups and provide insight into disease-specific factors influencing motor recovery potential.

Previous tDCS studies have found significant results with sample sizes between 10-20 participants for a two-round study comparing training sessions with real tDCS versus sessions done without tDCS. However, the investigators plan to recruit 30 participants living with each condition as this will allow us to examine results per group, but also how the individual groups compare.

ELIGIBILITY:
Inclusion Criteria:

- 1. Participants must be able to walk unassisted, or with the assistance of a walker or cane, and be individuals who walk daily.

2. Participants should have a sufficient level of English to be able to express themselves verbally, be able to read and follow instructions.

Exclusion Criteria:

* 3. Individuals with metal implants within the brain such as shunts will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Gait speed | Measures collected at three points each round: baseline in week 1, post-treatment at the final stimulation session, and follow-up two weeks after the final session.
  Within each round, scores from the final week and final session of real tDCS stimulation will be compared to performance during the first week and final sham tDCS session to check for significant improvement. Our primary outcome measures will be those found for gait; for example, a faster walking time subsequent to tDCS stimulation compared to the placebo baseline. Participants will also return two weeks later for a post-stimulation evaluation to check if improvement was maintained. To check if the arrangement of electrodes impacts the effect, times from the final tDCS session of each round will be compared.

SECONDARY OUTCOMES:
Articulation Quality (Clinician-Rated Speech Production on Word and Sentence Repetition) | Measures collected at three points each round: baseline in week 1, post-treatment at the final stimulation session, and follow-up two weeks after the final session.
  Articulation will be assessed using a clinician-administered repetition task involving single words and short sentences. Speech production quality will be rated by the clinician using a standardized 5-point articulation quality scale (1 = severely distorted, 5 = normal/near-normal production). The reported value will be the rating score.
Eye-Gaze Control (Clinician-Rated Ability to Track a Moving Target) | Measures collected at three points each round: baseline in week 1, post-treatment at the final stimulation session, and follow-up two weeks after the final session.
  Eye-gaze performance will be evaluated using a bedside oculomotor task. Participants are asked to follow a moving pencil with their eyes while keeping their head still. A clinician will rate eye-gaze control on a standardized 3-point scale (0 = unable, 1 = inconsistent, 2 = consistent and accurate). The reported value will be the rating score.

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Roncero, Ph.D, Principal Investigator — Baycrest Academy of Health Sciences and Geriatric Research; Howard Chertkow, MD, Principal Investigator — Baycrest Academy of Health Sciences and Geriatric Research
Locations (1):
- Baycrest Academy of Health Sciences and Geriatric Research, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Only aggregated, de-identified summary results will be made available through publications, presentations, or upon request.

DOCUMENTS (1):
  • Study Protocol (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT07291687/Prot_000.pdf